CLINICAL TRIAL: NCT03832621
Title: NIVOLUMAB Plus IPILIMUMAB and TEMOZOLOMIDE in Combination in Microsatellite Stable (MSS), MGMT Silenced Metastatic Colorectal Cancer (mCRC): the MAYA Study
Brief Title: NIVOLUMAB Plus IPILIMUMAB and TEMOZOLOMIDE in Microsatellite Stable, MGMT Silenced Metastatic Colorectal Cancer
Acronym: MAYA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT202-18
Record Dates: First submitted 2019-01-31; First posted 2019-02-06 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: nivolumab; ipilimumab; temozolomide; microsatellite stable; MSS; MGMT
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Temozolomide; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- temozolomide + nivolumab + ipilimumab (Experimental): Temozolomide 150 mg/sqm daily on days 1-5 every 4 weeks, for two cycles followed by TC scan assessment: if SD/PR/CR second treatment phase with nivolumab 480 mg i.v. every 4 weeks, low-dose ipilimumab 1 mg/Kg i.v. every 8 weeks and temozolomide at the previously adopted schedule
  Interventions: Drug: Temozolomide; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Temozolomide — temozolomide 150 mg/sqm daily on days 1-5 every 4 weeks
Drug: Nivolumab — nivolumab 480 mg i.v. every 4 weeks
Drug: Ipilimumab — low-dose ipilimumab 1 mg/Kg i.v. every 8 weeks

SUMMARY:
This is a Phase II, multicenter, single-arm trial designed to evaluate the efficacy and safety of nivolumab (NIVO), ipilimumab (IPI) and temozolomide (TMZ) combination in 27 patients with MSS, MGMT-silenced mCRC with initial clinical benefit following lead-in treatment with single-agent TMZ.

Immune checkpoint inhibitors have been shown to trigger durable antitumor effects in a subset of patients. A high number of tumor mutations (so called 'tumor mutational burden') has recently been found associated with increased immunogenicity (due to a high number of neoantigens) and improved treatment efficacy across several different solid tumors. In mCRCs, only a small fraction of tumors (<5%) display a high mutational load and are usually associated with inactivation of mismatch repair genes such as MLH1, MSH2 and MSH6. Checkpoint inhibitors may have increased activity in dMMR/microsatellite instability-high (MSI-H) tumors, a hypothesis which was tested in various Phase II trials with positive results. On the opposite, mismatch repair proficient colorectal cancer is unresponsive to immune checkpoint inhibitors.

Previous reports indicate that acquired resistance to TMZ may emerge through the induction of a microsatellite-instability-positive phenotype and recent data showed that inactivation of MMR, driven by acquired resistance to the clinical agent temozolomide, increased mutational load, promoted continuous renewal of neoantigens in human colorectal cancers and triggered immune surveillance in mouse models.

On all of the above grounds, the investigators hypothesize that treatment of microsatellite stable MGMT hypermethylated CRCs with alkylating agents could reshape the tumor genetic landscape by increasing the tumor mutational burden, leading to achieve potential sensitization to immunotherapy.

DETAILED DESCRIPTION:
In advanced CRC, the occurrence of chemorefractory disease poses a major therapeutic challenge for presence of an adequate performance status to potentially receive further treatments. Patients who progress after all approved treatments may be generally considered suitable for new investigational drugs or strategies. Thus, in the era of personalized medicine, tumor molecular profiling may lead to the identification of therapeutic targets or predictive biomarkers for pharmacological intervention. The DNA repair gene O6-methylguanine-DNA methyltransferase (MGMT) is responsible of the elimination of alkyl groups from the O6-position of guanine. If inactive, it may be involved in early steps of colorectal tumor genesis leading to an increase of G-to-A point mutations. Epigenetic silencing of MGMT during colorectal tumor genesis is associated with hypermethylation of the CpG island in its promoter. This transcriptional gene silencing is responsible for diminished DNA-repair of O6-alkylguanine adducts, with the consequence of enhancing chemosensitivity to alkylating agents including dacarbazine and its oral prodrug temozolomide (TMZ). Previous phase II studies showed that TMZ induced an average objective response rate by RECIST criteria in 10% of heavily pre-treated patients with advanced CRC carrying MGMT promoter methylated tumors. Thus, MGMT methylation by methylation-specific PCR (MSP) used for patients screening seemed to be a necessary but not sufficient condition to identify response to TMZ. Digital PCR quantification of MGMT methylation refined patients' selection, with benefit restricted to those with highly hyper-methylated tumors. Further analysis showed that MGMT negative/low expression by immunohistochemistry (IHC) is found in about one third of MSP-methylated samples and is associated with increased response rate. However, even in responding mCRC patients, acquired resistance to single agent TMZ emerges rapidly and almost invariably within 6 months from treatment initiation.

Immune checkpoint inhibitors have been shown to trigger durable antitumor effects in a subset of patients. A high number of tumor mutations (so called 'tumor mutational burden') has recently been found associated with increased immunogenicity (due to a high number of neoantigens) and improved treatment efficacy across several different solid tumors. Early clinical testing indicated that only 1 of 33 CRC patients had a response to anti PD-1 treatment, in contrast to substantial fractions of patients with melanomas, renal-cell cancers, and lung tumors who showed benefit from PD-1 blockade. Similarly, anti CTLA-4 treatment up today brought to unsatisfactory results in unselected mCRC patients. The probability of response has been ascribed to a high mutational burden (that is an elevated number of somatic mutations), which translates in increased number of neo-antigens. In mCRCs, only a small fraction of tumors (<5%) display a high mutational load and are usually associated with inactivation of mismatch repair genes such as MLH1, MSH2 and MSH6. Molecular alterations in these genes occur as an initial step in colon tumor genesis leading to the microsatellite instability (MSI) phenotype. Indeed, mismatch repair-deficient (dMMR) colorectal cancers have 10 to 100 times as many somatic mutations as mismatch repair-proficient colorectal cancers. Moreover, mismatch repair-deficient cancers contain prominent lymphocyte infiltrates, a finding consistent with an immune response. Thus, checkpoint inhibitors may have increased activity in dMMR/microsatellite instability-high (MSI-H) tumors, a hypothesis which was tested in various Phase II trials with positive results. On the opposite, mismatch repair proficient colorectal cancer is unresponsive to immune checkpoint inhibitors.

Previous reports indicate that acquired resistance to TMZ may emerge through the induction of a microsatellite-instability-positive phenotype. On the other hand, TMZ by itself has been shown to induce an increase of mutational load in other MGMT deficient solid tumors such as melanoma or glioblastoma. In parallel, other studies have demonstrated that alkylating agents' side effects can influence the immune cell compartment by selectively depleting the immuno-suppressive T regulator lymphocytes (Tregs), and activating the immuno-active T cytotoxic lymphocytes (Tc) and natural killers (NK). The investigators recently showed that inactivation of MMR, driven by acquired resistance to the clinical agent temozolomide, increased mutational load, promoted continuous renewal of neoantigens in human colorectal cancers and triggered immune surveillance in mouse models.

On all of the above grounds, the investigators hypothesize that treatment of microsatellite stable MGMT hypermethylated CRCs with alkylating agents could reshape the tumor genetic landscape by increasing the tumor mutational burden either directly (by inducing G>A mutations) or/and indirectly (by inactivating DNA repair genes such as MLH1, MSH2 or MSH6, which in turn could lead to hypermutated phenotype) therefore enhancing formation of cancer neoantigens and immunogenicity. TMZ treatment can also modulate the repertoire of immune cells (Tregs, Tc, NK) favoring T cell activation. To achieve potential sensitization to immunotherapy by means of TMZ-induced MSI-like status, treatment with TMZ should be active (i.e. inducing a SD/PR/CR).

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent prior to any study specific procedures
2. Willing and able to comply with the protocol
3. ≥18 years of age
4. ECOG status 0 - 1
5. At least 12 weeks of life expectancy at time of entry into the study
6. Histologically confirmed metastatic or inoperable adenocarcinoma of the colon and/or rectum, with centrally confirmed mismatch repair proficiency (microsatellite stable [MSS]) by multiplex polymerase chain reaction (PCR), MGMT promoter methylation by methylation-specific PCR (MSP) and MGMT low expression by IHC
7. Patients with progressive disease or that are not candidate for oxaliplatin irinotecan fluoropirimidin based chemotherapy and anti EGFR mAbs (in RAS/BRAF wild type tumors) in the metastatic setting
8. Patients with documented disease relapsed within 6 months from the completion of adjuvant oxaliplatin-based chemotherapy are considered eligible
9. Measureable, unresectable disease according to RECIST 1.1. Subjects with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll provided the lesion(s) have demonstrated clear progression and can be measured accurately.
10. Is willing and able to provide an adequate archival tumor sample (FFPE) available for tissue screening for central tissue screening. If the tumour block is not available, a minimum of twenty 3-micron unstained sections on charged slides of tumor will be required.

Exclusion Criteria:

1. Requirement for treatment with any medicinal product that contraindicates the use of any of the study medications, may interfere with the planned treatment, affects patient compliance or puts the patient at high risk for treatment-related complications
2. Inability to swallow pills
3. Refractory nausea and vomiting, malabsorption, external biliary shunt or significant bowel resection that would preclude adequate absorption
4. Inadequate haematological function indicated by all of the following:

   * White Blood Cell (WBC) count < 2 x 109/L
   * Absolute neutrophil count (ANC) < 1.5 x 109/L
   * Platelet count < 100 x 109/L
   * Haemoglobin < 9 g/dL (patients may have transfusions and/or growth factors to attain adequate Hb)
5. Inadequate liver function indicated by all of the following:

   * Total bilirubin ≥ 1.5 x upper limit of normal (ULN)
   * Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≥ 3 x ULN (≥ 5 x ULN in patients with known liver metastases)
   * Alkaline phosphatase (ALP) ≥ 2 x ULN (≥ 5 x ULN in patients with known liver metastases)
6. Inadequate renal function indicated by all of the following:

   - Serum creatinine > 1.5 x ULN or calculated creatinine clearance < 40 ml/min
7. INR > 1.5 and aPTT > 1.5 x ULN within 7 days prior to the start of study treatment for patients not receiving anti-coagulation

   a. NOTE: The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least two weeks prior to the start of study treatment
8. Active infection requiring intravenous antibiotics at the start of study treatment
9. Previous or concurrent malignancy, except for adequately treated basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast, or other cancer for which the patient has been disease-free for three years prior to study entry
10. Evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any of the study medications, puts the patient at higher risk for treatment-related complications or may affect the interpretation of study results
11. Clinically significant (i.e. active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to start of study treatment, myocardial infarction ≤ 6 months prior to study enrolment, unstable angina, New York Heart Association (NYHA) Functional Classification Grade II or greater congestive heart failure, or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
12. History or evidence upon physical or neurological examination of central nervous system (CNS) disease (e.g. seizures) unrelated to cancer unless adequately treated with standard medical therapy
13. Active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI except where contraindicated in which CT scan is acceptable) evidence of progression for at least 8 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. Cases should be discussed with the medical monitor. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (>10mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
14. Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to start of study treatment, or anticipation of need for major surgical procedure during the course of the study.
15. Treatment with any chemotherapy, curative intent radiation therapy, biologics for cancer, or investigational therapy within 28 days of first administration of study treatment (subjects with prior cytotoxic or investigational products < 4 weeks prior to treatment might be eligible after discussion between investigator and sponsor, if toxicities from the prior treatment have been resolved to Grade 1 (NCI CTCAE version 4). Prior focal palliative radiotherapy must have been completed at least 2 weeks before study drug administration.
16. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 4) or baseline before administration of study drug. Subjects with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum based therapy, are permitted to enroll.
17. Known hypersensitivity to any of the study medications or Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of the NIVO formulation
18. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
19. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis (see Appendix IV for a more comprehensive list of autoimmune diseases)

    a. Note: history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible. Subjects with controlled type I diabetes mellitus on a stable insulin regimen, vitiligo or psoriasis not requiring systemic treatment may be eligible.
20. Prior allogeneic bone marrow transplantation or prior solid organ transplantation
21. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on Screening chest CT scan
22. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to start of study treatment
23. Treatment with systemic corticosteroids (>10 mg daily prednisone equivalents) or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor [TNF] agents) within 2 weeks prior to start of study treatment, or requirement for systemic immunosuppressive medications during the trial. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.

    a. Note: Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the Sponsor.
24. Positive test for human immunodeficiency virus (HIV)
25. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test prior to randomization) or hepatitis C

    1. Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible. Patients with detectable HBV-DNA are not eligible.
    2. Note: Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid (RNA).
26. Active tuberculosis
27. Administration of a live, attenuated vaccine within 4 weeks prior to start of study treatment or anticipation that such a live attenuated vaccine will be required during the study
28. Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including prior therapy with anti-tumor vaccines.
29. Pregnancy or lactation. A serum pregnancy test is required within 7 days prior to start of study treatment, or within 14 days with a confirmatory urine pregnancy test within 7 days prior start of study treatment
30. For women who are not post-menopausal (< 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): refusal to use a highly effective contraceptive method (i.e. with a failure rate of < 1% per year such as sexual abstinence, hormonal implants, combined oral contraceptives, vasectomised partner), during the study drug administration and for at least 6 months after the last dose of study medication. Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception. A combination of male condom with cap, diaphragm or sponge with spermicide (double barrier methods) is not considered highly effective, birth control methods. Acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. A Vasectomised partner is a highly effective birth control method provided that partner is the sole sexual partner of the trial participant and that the vasectomised partner has received medical assessment of the surgical success.
31. For men: refusal to use a highly effective contraceptive method (i.e. with a failure rate of < 1 % per year such as vasectomy, sexual abstinence or female partner use of hormonal implants or combined oral contraceptives) during the study drug administration and for a period of at least 6 months after the last dose of study medication. Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable methods of contraception. A combination of male condom with either, cap, diaphragm or sponge with spermicide (double barrier methods) is not considered highly effective, birth control methods. Acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. A vasectomised trial participant is a highly effective birth control method provided that the trial participant has received medical assessment of the surgical success.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy, measured as 8-month PFS rate, of the combination of temozolomide, nivolumab and ipilimumab in patients achieving disease control following 2-month lead-in treatment with single agent TMZ | 8 months from the last patient enrolled
  The primary efficacy endpoint of this study is 8-month PFS rate, defined as the proportion of patients alive and progression-free at 8 months from the enrollment.
  Investigator-assessed PFS according to RECIST v1.1 Investigator-assessed PFS according to modified RECIST

SECONDARY OUTCOMES:
Estimate the overall response rates (ORR) of the combination regimen of temozolomide, nivolumab and ipilimumab | 36 months
  ORR measured by response rate according to RECIST 1.1 and modified RECIST criteria
Estimate duration of response (DoR) of the combination regimen of temozolomide, nivolumab and ipilimumab | 36 months
  DoR assessed per RECIST 1.1 and modified RECIST
Estimate overall survival (OS) of the combination regimen of temozolomide, nivolumab and ipilimumab | 36 months
  overall survival
Estimate ORR according to an Imaging Independent Central Review, using RECIST 1.1 and modified RECIST criteria | 36 moths
  CD-ROM copies of the CT scans performed at baseline and during treatment until disease progression according to RECIST 1.1 and modified RECIST criteria will be collected at the Coordinating Center (S.C. Oncologia Medica 1, Fondazione IRCCS Istituto Nazionale dei Tumori) for central review
Evaluate the adverse events encountered by patients treated with the combination of temozolomide, nivolumab and ipilimumab | 36 months
  Number of participants with treatment-related adverse events graded according to the NCI CTCAE v4.0
Estimate DoR of the combination regimen of temozolomide, nivolumab and ipilimumab according to an Imaging Independent Central Review | 36 months
  DoR calculated after the Imaging Independent Central Review
Estimate PFS of the combination regimen of temozolomide, nivolumab and ipilimumab according to an Imaging Independent Central Review | 36 months
  PFS calculated after the Imaging Independent Central Review
Assess quality of life | 36 months
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. PRO will be assessed by EORTC QLQ-C30 EORTC QLQ-CR29 and EuroQol EQ-5D

OTHER OUTCOMES:
Evaluate the relationship between tumor and plasma MGMT methylation | 36 months
  Quantification of the percentage of MGMT methylation with digital PCR for MGMT methylation status will be performed in archival tumor tissue, tumor re-biopsies and cell-free circulating DNA (cfDNA) (cfDNA)
Evaluate the tumor mutational load | 36 months
  Mutational load will be assessed in archival tumor tissues, tumor biopsies and cfDNA by means of whole exome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Pietrantonio, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI, Italy

REFERENCES:
- [Background] Schmoll HJ, Van Cutsem E, Stein A, Valentini V, Glimelius B, Haustermans K, Nordlinger B, van de Velde CJ, Balmana J, Regula J, Nagtegaal ID, Beets-Tan RG, Arnold D, Ciardiello F, Hoff P, Kerr D, Kohne CH, Labianca R, Price T, Scheithauer W, Sobrero A, Tabernero J, Aderka D, Barroso S, Bodoky G, Douillard JY, El Ghazaly H, Gallardo J, Garin A, Glynne-Jones R, Jordan K, Meshcheryakov A, Papamichail D, Pfeiffer P, Souglakos I, Turhal S, Cervantes A. ESMO Consensus Guidelines for management of patients with colon and rectal cancer. a personalized approach to clinical decision making. Ann Oncol. 2012 Oct;23(10):2479-2516. doi: 10.1093/annonc/mds236. PMID 23012255
- [Background] Temraz S, Mukherji D, Shamseddine A. Sequencing of treatment in metastatic colorectal cancer: where to fit the target. World J Gastroenterol. 2014 Feb 28;20(8):1993-2004. doi: 10.3748/wjg.v20.i8.1993. PMID 24616571
- [Background] Stein A, Bokemeyer C. How to select the optimal treatment for first line metastatic colorectal cancer. World J Gastroenterol. 2014 Jan 28;20(4):899-907. doi: 10.3748/wjg.v20.i4.899. PMID 24574764
- [Background] Tejpar S, Piessevaux H. Personalized medicine in metastatic colorectal cancer treated with anti-epidermal growth factor receptor agents: a future opportunity? Asia Pac J Clin Oncol. 2014 Mar;10 Suppl 1:2-10. doi: 10.1111/ajco.12176. PMID 24512508
- [Background] Bekaii-Saab T, Wu C. Seeing the forest through the trees: a systematic review of the safety and efficacy of combination chemotherapies used in the treatment of metastatic colorectal cancer. Crit Rev Oncol Hematol. 2014 Jul;91(1):9-34. doi: 10.1016/j.critrevonc.2014.01.001. Epub 2014 Jan 15. PMID 24534706
- [Background] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Background] Mayer RJ, Van Cutsem E, Falcone A, Yoshino T, Garcia-Carbonero R, Mizunuma N, Yamazaki K, Shimada Y, Tabernero J, Komatsu Y, Sobrero A, Boucher E, Peeters M, Tran B, Lenz HJ, Zaniboni A, Hochster H, Cleary JM, Prenen H, Benedetti F, Mizuguchi H, Makris L, Ito M, Ohtsu A; RECOURSE Study Group. Randomized trial of TAS-102 for refractory metastatic colorectal cancer. N Engl J Med. 2015 May 14;372(20):1909-19. doi: 10.1056/NEJMoa1414325. PMID 25970050
- [Background] Oberg A, Samii S, Stenling R, Lindmark G. Different occurrence of CD8+, CD45R0+, and CD68+ immune cells in regional lymph node metastases from colorectal cancer as potential prognostic predictors. Int J Colorectal Dis. 2002 Jan;17(1):25-9. doi: 10.1007/s003840100337. PMID 12018450
- [Background] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Background] Pages F, Kirilovsky A, Mlecnik B, Asslaber M, Tosolini M, Bindea G, Lagorce C, Wind P, Marliot F, Bruneval P, Zatloukal K, Trajanoski Z, Berger A, Fridman WH, Galon J. In situ cytotoxic and memory T cells predict outcome in patients with early-stage colorectal cancer. J Clin Oncol. 2009 Dec 10;27(35):5944-51. doi: 10.1200/JCO.2008.19.6147. Epub 2009 Oct 26. PMID 19858404
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Ribas A, Puzanov I, Dummer R, Schadendorf D, Hamid O, Robert C, Hodi FS, Schachter J, Pavlick AC, Lewis KD, Cranmer LD, Blank CU, O'Day SJ, Ascierto PA, Salama AK, Margolin KA, Loquai C, Eigentler TK, Gangadhar TC, Carlino MS, Agarwala SS, Moschos SJ, Sosman JA, Goldinger SM, Shapira-Frommer R, Gonzalez R, Kirkwood JM, Wolchok JD, Eggermont A, Li XN, Zhou W, Zernhelt AM, Lis J, Ebbinghaus S, Kang SP, Daud A. Pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory melanoma (KEYNOTE-002): a randomised, controlled, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):908-18. doi: 10.1016/S1470-2045(15)00083-2. Epub 2015 Jun 23. PMID 26115796
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Lipson EJ, Sharfman WH, Drake CG, Wollner I, Taube JM, Anders RA, Xu H, Yao S, Pons A, Chen L, Pardoll DM, Brahmer JR, Topalian SL. Durable cancer regression off-treatment and effective reinduction therapy with an anti-PD-1 antibody. Clin Cancer Res. 2013 Jan 15;19(2):462-8. doi: 10.1158/1078-0432.CCR-12-2625. Epub 2012 Nov 20. PMID 23169436
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Goldstein J, Tran B, Ensor J, Gibbs P, Wong HL, Wong SF, Vilar E, Tie J, Broaddus R, Kopetz S, Desai J, Overman MJ. Multicenter retrospective analysis of metastatic colorectal cancer (CRC) with high-level microsatellite instability (MSI-H). Ann Oncol. 2014 May;25(5):1032-8. doi: 10.1093/annonc/mdu100. Epub 2014 Feb 27. PMID 24585723
- [Background] Koopman M, Kortman GA, Mekenkamp L, Ligtenberg MJ, Hoogerbrugge N, Antonini NF, Punt CJ, van Krieken JH. Deficient mismatch repair system in patients with sporadic advanced colorectal cancer. Br J Cancer. 2009 Jan 27;100(2):266-73. doi: 10.1038/sj.bjc.6604867. PMID 19165197
- [Background] Segal NH, Parsons DW, Peggs KS, Velculescu V, Kinzler KW, Vogelstein B, Allison JP. Epitope landscape in breast and colorectal cancer. Cancer Res. 2008 Feb 1;68(3):889-92. doi: 10.1158/0008-5472.CAN-07-3095. PMID 18245491
- [Background] Cancer Genome Atlas Network. Comprehensive molecular characterization of human colon and rectal cancer. Nature. 2012 Jul 18;487(7407):330-7. doi: 10.1038/nature11252. PMID 22810696
- [Background] Timmermann B, Kerick M, Roehr C, Fischer A, Isau M, Boerno ST, Wunderlich A, Barmeyer C, Seemann P, Koenig J, Lappe M, Kuss AW, Garshasbi M, Bertram L, Trappe K, Werber M, Herrmann BG, Zatloukal K, Lehrach H, Schweiger MR. Somatic mutation profiles of MSI and MSS colorectal cancer identified by whole exome next generation sequencing and bioinformatics analysis. PLoS One. 2010 Dec 22;5(12):e15661. doi: 10.1371/journal.pone.0015661. PMID 21203531
- [Background] Smyrk TC, Watson P, Kaul K, Lynch HT. Tumor-infiltrating lymphocytes are a marker for microsatellite instability in colorectal carcinoma. Cancer. 2001 Jun 15;91(12):2417-22. PMID 11413533
- [Background] Overman MJ, McDermott R, Leach JL, Lonardi S, Lenz HJ, Morse MA, Desai J, Hill A, Axelson M, Moss RA, Goldberg MV, Cao ZA, Ledeine JM, Maglinte GA, Kopetz S, Andre T. Nivolumab in patients with metastatic DNA mismatch repair-deficient or microsatellite instability-high colorectal cancer (CheckMate 142): an open-label, multicentre, phase 2 study. Lancet Oncol. 2017 Sep;18(9):1182-1191. doi: 10.1016/S1470-2045(17)30422-9. Epub 2017 Jul 19. PMID 28734759
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Esteller M, Herman JG. Generating mutations but providing chemosensitivity: the role of O6-methylguanine DNA methyltransferase in human cancer. Oncogene. 2004 Jan 8;23(1):1-8. doi: 10.1038/sj.onc.1207316. PMID 14712205
- [Background] Ju HX, An B, Okamoto Y, Shinjo K, Kanemitsu Y, Komori K, Hirai T, Shimizu Y, Sano T, Sawaki A, Tajika M, Yamao K, Fujii M, Murakami H, Osada H, Ito H, Takeuchi I, Sekido Y, Kondo Y. Distinct profiles of epigenetic evolution between colorectal cancers with and without metastasis. Am J Pathol. 2011 Apr;178(4):1835-46. doi: 10.1016/j.ajpath.2010.12.045. Epub 2011 Mar 4. PMID 21406167
- [Background] Barault L, Amatu A, Bleeker FE, Moutinho C, Falcomata C, Fiano V, Cassingena A, Siravegna G, Milione M, Cassoni P, De Braud F, Ruda R, Soffietti R, Venesio T, Bardelli A, Wesseling P, de Witt Hamer P, Pietrantonio F, Siena S, Esteller M, Sartore-Bianchi A, Di Nicolantonio F. Digital PCR quantification of MGMT methylation refines prediction of clinical benefit from alkylating agents in glioblastoma and metastatic colorectal cancer. Ann Oncol. 2015 Sep;26(9):1994-1999. doi: 10.1093/annonc/mdv272. Epub 2015 Jun 25. PMID 26113646
- [Background] Shima K, Morikawa T, Baba Y, Nosho K, Suzuki M, Yamauchi M, Hayashi M, Giovannucci E, Fuchs CS, Ogino S. MGMT promoter methylation, loss of expression and prognosis in 855 colorectal cancers. Cancer Causes Control. 2011 Feb;22(2):301-9. doi: 10.1007/s10552-010-9698-z. Epub 2010 Dec 8. PMID 21140203
- [Background] Amatu A, Sartore-Bianchi A, Moutinho C, Belotti A, Bencardino K, Chirico G, Cassingena A, Rusconi F, Esposito A, Nichelatti M, Esteller M, Siena S. Promoter CpG island hypermethylation of the DNA repair enzyme MGMT predicts clinical response to dacarbazine in a phase II study for metastatic colorectal cancer. Clin Cancer Res. 2013 Apr 15;19(8):2265-72. doi: 10.1158/1078-0432.CCR-12-3518. Epub 2013 Feb 19. PMID 23422094
- [Background] Hochhauser D, Glynne-Jones R, Potter V, Gravalos C, Doyle TJ, Pathiraja K, Zhang Q, Zhang L, Sausville EA. A phase II study of temozolomide in patients with advanced aerodigestive tract and colorectal cancers and methylation of the O6-methylguanine-DNA methyltransferase promoter. Mol Cancer Ther. 2013 May;12(5):809-18. doi: 10.1158/1535-7163.MCT-12-0710. Epub 2013 Feb 26. PMID 23443801
- [Background] Pietrantonio F, Perrone F, de Braud F, Castano A, Maggi C, Bossi I, Gevorgyan A, Biondani P, Pacifici M, Busico A, Gariboldi M, Festinese F, Tamborini E, Di Bartolomeo M. Activity of temozolomide in patients with advanced chemorefractory colorectal cancer and MGMT promoter methylation. Ann Oncol. 2014 Feb;25(2):404-8. doi: 10.1093/annonc/mdt547. Epub 2013 Dec 29. PMID 24379162
- [Background] Bardelli A, Cahill DP, Lederer G, Speicher MR, Kinzler KW, Vogelstein B, Lengauer C. Carcinogen-specific induction of genetic instability. Proc Natl Acad Sci U S A. 2001 May 8;98(10):5770-5. doi: 10.1073/pnas.081082898. Epub 2001 Apr 10. PMID 11296254
- [Background] Yip S, Miao J, Cahill DP, Iafrate AJ, Aldape K, Nutt CL, Louis DN. MSH6 mutations arise in glioblastomas during temozolomide therapy and mediate temozolomide resistance. Clin Cancer Res. 2009 Jul 15;15(14):4622-9. doi: 10.1158/1078-0432.CCR-08-3012. Epub 2009 Jul 7. PMID 19584161
- [Background] Alexandrov LB, Jones PH, Wedge DC, Sale JE, Campbell PJ, Nik-Zainal S, Stratton MR. Clock-like mutational processes in human somatic cells. Nat Genet. 2015 Dec;47(12):1402-7. doi: 10.1038/ng.3441. Epub 2015 Nov 9. PMID 26551669
- [Background] Su YB, Sohn S, Krown SE, Livingston PO, Wolchok JD, Quinn C, Williams L, Foster T, Sepkowitz KA, Chapman PB. Selective CD4+ lymphopenia in melanoma patients treated with temozolomide: a toxicity with therapeutic implications. J Clin Oncol. 2004 Feb 15;22(4):610-6. doi: 10.1200/JCO.2004.07.060. Epub 2004 Jan 15. PMID 14726505
- [Background] Hervieu A, Rebe C, Vegran F, Chalmin F, Bruchard M, Vabres P, Apetoh L, Ghiringhelli F, Mignot G. Dacarbazine-mediated upregulation of NKG2D ligands on tumor cells activates NK and CD8 T cells and restrains melanoma growth. J Invest Dermatol. 2013 Feb;133(2):499-508. doi: 10.1038/jid.2012.273. Epub 2012 Sep 6. PMID 22951720
- [Background] Fritzell S, Sanden E, Eberstal S, Visse E, Darabi A, Siesjo P. Intratumoral temozolomide synergizes with immunotherapy in a T cell-dependent fashion. Cancer Immunol Immunother. 2013 Sep;62(9):1463-74. doi: 10.1007/s00262-013-1449-z. Epub 2013 Jun 18. PMID 23775421
- [Background] Sharpe AH, Wherry EJ, Ahmed R, Freeman GJ. The function of programmed cell death 1 and its ligands in regulating autoimmunity and infection. Nat Immunol. 2007 Mar;8(3):239-45. doi: 10.1038/ni1443. PMID 17304234
- [Background] Robert C, Thomas L, Bondarenko I, O'Day S, Weber J, Garbe C, Lebbe C, Baurain JF, Testori A, Grob JJ, Davidson N, Richards J, Maio M, Hauschild A, Miller WH Jr, Gascon P, Lotem M, Harmankaya K, Ibrahim R, Francis S, Chen TT, Humphrey R, Hoos A, Wolchok JD. Ipilimumab plus dacarbazine for previously untreated metastatic melanoma. N Engl J Med. 2011 Jun 30;364(26):2517-26. doi: 10.1056/NEJMoa1104621. Epub 2011 Jun 5. PMID 21639810
- [Background] Pietrantonio F, de Braud F, Milione M, Maggi C, Iacovelli R, Dotti KF, Perrone F, Tamborini E, Caporale M, Berenato R, Leone G, Pellegrinelli A, Bossi I, Festinese F, Federici S, Di Bartolomeo M. Dose-Dense Temozolomide in Patients with MGMT-Silenced Chemorefractory Colorectal Cancer. Target Oncol. 2016 Jun;11(3):337-43. doi: 10.1007/s11523-015-0397-2. PMID 26538496
- [Background] Calegari MA, Inno A, Monterisi S, Orlandi A, Santini D, Basso M, Cassano A, Martini M, Cenci T, de Pascalis I, Camarda F, Barbaro B, Larocca LM, Gori S, Tonini G, Barone C. A phase 2 study of temozolomide in pretreated metastatic colorectal cancer with MGMT promoter methylation. Br J Cancer. 2017 May 9;116(10):1279-1286. doi: 10.1038/bjc.2017.109. Epub 2017 Apr 20. PMID 28427088
- [Background] Tosolini M, Kirilovsky A, Mlecnik B, Fredriksen T, Mauger S, Bindea G, Berger A, Bruneval P, Fridman WH, Pages F, Galon J. Clinical impact of different classes of infiltrating T cytotoxic and helper cells (Th1, th2, treg, th17) in patients with colorectal cancer. Cancer Res. 2011 Feb 15;71(4):1263-71. doi: 10.1158/0008-5472.CAN-10-2907. Epub 2011 Feb 8. PMID 21303976
- [Background] Deaglio S, Mehta K, Malavasi F. Human CD38: a (r)evolutionary story of enzymes and receptors. Leuk Res. 2001 Jan;25(1):1-12. doi: 10.1016/s0145-2126(00)00093-x. PMID 11137554
- [Background] Vaisitti T, Aydin S, Rossi D, Cottino F, Bergui L, D'Arena G, Bonello L, Horenstein AL, Brennan P, Pepper C, Gaidano G, Malavasi F, Deaglio S. CD38 increases CXCL12-mediated signals and homing of chronic lymphocytic leukemia cells. Leukemia. 2010 May;24(5):958-69. doi: 10.1038/leu.2010.36. Epub 2010 Mar 11. PMID 20220774
- [Background] Malavasi F, Deaglio S, Damle R, Cutrona G, Ferrarini M, Chiorazzi N. CD38 and chronic lymphocytic leukemia: a decade later. Blood. 2011 Sep 29;118(13):3470-8. doi: 10.1182/blood-2011-06-275610. Epub 2011 Jul 15. PMID 21765022
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Pennock GK, Waterfield W, Wolchok JD. Patient responses to ipilimumab, a novel immunopotentiator for metastatic melanoma: how different are these from conventional treatment responses? Am J Clin Oncol. 2012 Dec;35(6):606-11. doi: 10.1097/COC.0b013e318209cda9. PMID 21336089
- [Background] Hoos A, Ibrahim R, Korman A, Abdallah K, Berman D, Shahabi V, Chin K, Canetta R, Humphrey R. Development of ipilimumab: contribution to a new paradigm for cancer immunotherapy. Semin Oncol. 2010 Oct;37(5):533-46. doi: 10.1053/j.seminoncol.2010.09.015. PMID 21074069
- [Background] Marventano S, Forjaz M, Grosso G, Mistretta A, Giorgianni G, Platania A, Gangi S, Basile F, Biondi A. Health related quality of life in colorectal cancer patients: state of the art. BMC Surg. 2013;13 Suppl 2(Suppl 2):S15. doi: 10.1186/1471-2482-13-S2-S15. Epub 2013 Oct 8. PMID 24267735
- [Background] Di Giacomo AM, Biagioli M, Maio M. The emerging toxicity profiles of anti-CTLA-4 antibodies across clinical indications. Semin Oncol. 2010 Oct;37(5):499-507. doi: 10.1053/j.seminoncol.2010.09.007. PMID 21074065
- [Background] Esteller M, Toyota M, Sanchez-Cespedes M, Capella G, Peinado MA, Watkins DN, Issa JP, Sidransky D, Baylin SB, Herman JG. Inactivation of the DNA repair gene O6-methylguanine-DNA methyltransferase by promoter hypermethylation is associated with G to A mutations in K-ras in colorectal tumorigenesis. Cancer Res. 2000 May 1;60(9):2368-71. PMID 10811111
- [Background] Oesch F, Klein S. Relevance of environmental alkylating agents to repair protein O6-alkylguanine-DNA alkyltransferase: determination of individual and collective repair capacities of O6-methylguanine. Cancer Res. 1992 Apr 1;52(7):1801-3. PMID 1532345
- [Background] Fehrenbacher L, Spira A, Ballinger M, Kowanetz M, Vansteenkiste J, Mazieres J, Park K, Smith D, Artal-Cortes A, Lewanski C, Braiteh F, Waterkamp D, He P, Zou W, Chen DS, Yi J, Sandler A, Rittmeyer A; POPLAR Study Group. Atezolizumab versus docetaxel for patients with previously treated non-small-cell lung cancer (POPLAR): a multicentre, open-label, phase 2 randomised controlled trial. Lancet. 2016 Apr 30;387(10030):1837-46. doi: 10.1016/S0140-6736(16)00587-0. Epub 2016 Mar 10. PMID 26970723
- [Background] Rosenberg JE, Hoffman-Censits J, Powles T, van der Heijden MS, Balar AV, Necchi A, Dawson N, O'Donnell PH, Balmanoukian A, Loriot Y, Srinivas S, Retz MM, Grivas P, Joseph RW, Galsky MD, Fleming MT, Petrylak DP, Perez-Gracia JL, Burris HA, Castellano D, Canil C, Bellmunt J, Bajorin D, Nickles D, Bourgon R, Frampton GM, Cui N, Mariathasan S, Abidoye O, Fine GD, Dreicer R. Atezolizumab in patients with locally advanced and metastatic urothelial carcinoma who have progressed following treatment with platinum-based chemotherapy: a single-arm, multicentre, phase 2 trial. Lancet. 2016 May 7;387(10031):1909-20. doi: 10.1016/S0140-6736(16)00561-4. Epub 2016 Mar 4. PMID 26952546
- [Derived] Morano F, Raimondi A, Pagani F, Lonardi S, Salvatore L, Cremolini C, Murgioni S, Randon G, Palermo F, Antonuzzo L, Pella N, Racca P, Prisciandaro M, Niger M, Corti F, Bergamo F, Zaniboni A, Ratti M, Palazzo M, Cagnazzo C, Calegari MA, Marmorino F, Capone I, Conca E, Busico A, Brich S, Tamborini E, Perrone F, Di Maio M, Milione M, Di Bartolomeo M, de Braud F, Pietrantonio F. Temozolomide Followed by Combination With Low-Dose Ipilimumab and Nivolumab in Patients With Microsatellite-Stable, O6-Methylguanine-DNA Methyltransferase-Silenced Metastatic Colorectal Cancer: The MAYA Trial. J Clin Oncol. 2022 May 10;40(14):1562-1573. doi: 10.1200/JCO.21.02583. Epub 2022 Mar 8. PMID 35258987